CLINICAL TRIAL: NCT03775096
Title: The Effect of Adrenergic Blocker Therapy on Cardiac and Striatal Transporter Uptake in Pre-Motor and Symptomatic Parkinson's Disease
Brief Title: Adrenergic Blockers for Cardiac Changes in Early Parkinson's Disease (Protocol 53136)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michele Tagliati, MD (Other)
Responsible Party: Sponsor-Investigator, Michele Tagliati, MD, Professor and Vice Chairman, Director of Movement Disorders, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1223-7784
Record Dates: First submitted 2018-12-09; First posted 2018-12-13 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-01

CONDITIONS: REM Sleep Behavior Disorder; Pre-motor Parkinson Disease; Symptomatic Parkinson Disease
Keywords: Early Parkinson Disease; REM Sleep Behaviour Disorder (RBD); carvedilol; Autonomic dysfunction; Neurodegeneration
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease, Secondary; Parkinson Disease; Primary Dysautonomias; Nerve Degeneration | interventions — Carvedilol

STUDY DESIGN:
Intervention Model Description: Treatment: carvedilol titration; Experimental treatment with carvedilol will be offered at stabilized medical treatment. The dosage of carvedilol will be gradually increased from the initial recommended starting dose of 3.125mg twice daily and will be doubled every week according to patient tolerability, as measured by subjective complaints, arterial blood pressure and heart rate. The target dose will be 25mg twice daily (50 mg/day). Subjects that cannot tolerate the 50 mg daily dose, will be offered to continue at the 25 mg daily dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- carvedilol therapy (Experimental): The dosage of carvedilol will be gradually increased from the initial recommended starting dose of 3.125 mg twice/daily, the target dose will be 25mg twice daily (50 mg/day) and participants will take 50 mg/day carvedilol for 6 months.Subjects that cannot tolerate the 50 mg daily dose, will be offered to continue at the 25 mg daily dose.
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — At the end of Baseline visit, carvedilol 3.125 twice daily will be initiated and maintained for 1 week, increased to 6.25twice daily (dispensed at week 1visit), to 12.5mg twice daily (dispensed at week 2) and a max dose of 25mg twice daily (dispensed at week 4 visit), as tolerated. A subject that cannot tolerate at least a 25 mg daily dose will be excluded from the study. Subjects that cannot tolerate the 50 mg daily dose, will be offered to continue at the 25 mg daily dose. The project will include a washout period at study end.
  Other Names: Coreg

SUMMARY:
REM Behavior Sleep Disorder (RBD) is a sleep disorder causing people to 'act out' their dreams. A high percentage of individuals with idiopathic RBD (iRBD) are known to develop conditions affecting the neurons in the brain such as Parkinson's disease (PD). Based on the increased risk to develop PD, individuals with iRBD are currently considered ideal candidates for therapies that can possibly protects brain cells, due to the critical window of opportunity to intervene early before brain cell loss progresses significantly.

Early changes of PD are associated with a number of symptoms including loss of smell, constipation, anxiety and depression. In addition, early heart and brain abnormalities can be visualized using specialized imaging techniques called 123I-MIBG myocardial scintigraphy (MIBG) and dopamine transporter (DAT) single photon emission computerized tomography (SPECT) respectively. The combined presence of certain symptoms and the use of these imaging techniques are considered early markers of PD in individuals with iRBD.

In other conditions, like heart failure, MIBG abnormalities are reversed by drugs able to block excessive adrenergic stimulation, known as beta-blockers. In this study the investigators want to learn about the effect of treatment with the beta-blocker carvedilol on MIBG abnormalities found in iRBD patients at risk to develop PD. The investigators believe that reversing the MIBG abnormality might prelude to a slowing of the neurodegenerative process. This drug is approved by the U.S. Food and Drug Administration (FDA) for congestive heart failure, hypertension and left ventricular dysfunction after myocardial infarction. However, carvedilol is not approved by the FDA in patients with iRBD at risk for PD. The available doses for this drug oral formulations are 3.125mg, 6.25mg, 12.5mg and 25mg.

Changes visualized with the MIBG imaging technique will be correlated to the presence and severity of neurological (i.e. tremors, stiffness, slow movements, walking difficulties) and other symptoms associated with PD (i.e. abnormal smell, constipation, depression, color vision abnormalities), as measured by specific clinical scales and exams.

DETAILED DESCRIPTION:
Idiopathic Parkinson's disease (PD) is a progressive neurodegenerative disorder of unknown etiology, characterized by bradykinesia (slowness of movements) associated with tremor at rest and/or muscle rigidity. PD is typically associated with a significant loss of dopaminergic neurons in the substantia nigra pars compacta(SNpc).The resulting nigro-striatal degeneration can be detected and quantified using a dopamine transporter (DAT) single photon emission computerized tomography (SPECT) imaging technique. This type of imaging, recently approved for clinical use in the United States, uses a labeled ligand (123I-Ioflupane) with high affinity to the DAT in the striatum. The amount of transporter, which plays a crucial role in the health of the presynaptic dopaminergic neurons, is then visualized by SPECT. 123I-Ioflupane uptake is reduced 50-70% in patients with early PD.

In addition to cardinal motor symptoms, PD is characterized by a large number of "non-motor" symptoms (NMS), which add to the overall morbidity burden. Importantly, non--motor features may precede the diagnosis of PD, sometimes by several years. They include autonomic (gastrointestinal dysfunction, cardiovascular dysfunction with orthostatic hypotension (OH), urinary and sexual dysfunction, and hyperhidrosis), sleep (impaired sleep initiation and maintenance, rapid eye movement behavior disorder (RBD), sleep apnea and excessive daytime sleepiness), sensory (pain, hyposmia, and visual dysfunction), and neuropsychiatric disturbances (anhedonia, apathy, anxiety, depression, panic attacks, dementia, and psychosis).

Among NMS, cardiac dysautonomia is a common feature of PD, manifesting in 30% of patients as orthostatic hypotension, a symptom that is correlated to disease duration and severity. Cardiac sympathetic innervation (CSI) is also affected in PD and other synucleinopathies. Lewy Body (LB) pathology, widely considered a marker of PD when detected in the SNpc, is also found in the sinoatrial nodal ganglion and myocardium of PD patients at autopsy. Despite the high prevalence of both conditions, the relationship between CSI impairment and cardiac dysautonomia is still poorly understood.

Iodine-123 meta-iodobenzylguanidine (123I-MIBG) is an inactive physiological analogue that mimics the kinetics of norepinephrine (NE) and competes with NE for active cardiac uptake into the postganglionic sympathetic nerve terminal, where it is stored into granules by NE transport proteins. 123I-MIBG myocardial scintigraphy, an accepted measure of CSI, is abnormal in PD patients, with a characteristic reduction of Heart/Mediastinum (H/M) ratio (early and late uptake) and an increased Washout Rate (WR). 123I-MIBG uptake impairment is specific to PD and other synucleinopathies and can be used to differentiate PD and dementia with Lewy bodies (DLB) from other disorders with similar neurological phenomenology such as multiple system atrophy (MSA), progressive supranuclear palsy (PSP) and corticobasal degeneration (CBD).

123I-MIBG uptake deficit in PD is attributed to cardiac sympathetic denervation, based on neuropathological studies using tyrosine hydroxylase (TH) immunostaining in epicardial nerves. There is evidence of alpha-synuclein aggregation in the epicardial nerve fascicles - the distal axons of the cardiac sympathetic nerve - in subjects with incidental Lewy Body Disease (ILBD) at stage 2 or 3 of Braak staging with preserved TH immunoreactive axons, suggesting a preliminary stage in the development of cardiac sympathetic denervation. However, while 123I-MIBG myocardial scintigraphy abnormalities have been correlated with pre-motor symptoms like RBD, hyposmia and constipation, there is no pathological evidence of cardiac sympathetic denervation in subjects with signs of 123I-MIBG myocardial scintigraphy abnormality and recognized pre-motor symptoms of PD. Finally, despite the specific association with PD diagnosis, the relationship between CSI impairment and nigrostriatal degeneration is poorly understood. Two studies found a strong correlation between nigrostriatal dopaminergic degeneration, as measured by 123I Ioflupane SPECT, and CSI impairment at different stages of disease. 123I-MIBG uptake deficits have been correlated with the progression of the disease.

Interestingly, CSI - and therefore 123I-MIBG cardiac uptake - is impaired in other chronic conditions such as Heart Failure (HF), Hypertension, Diabetes Mellitus, Chronic Obstructive Pulmonary Disease and Sleep Apnea, with an identical pattern of abnormality as the one detected in PD patients. As opposed to cardiac sympathetic denervation, 123I-MIBG cardiac uptake impairment in these chronic conditions - and in particular HF - is explained with the hyperactivity of the sympathetic nervous system (SNS) acting as compensatory mechanism related to specific organ failure (i.e. post-ischemic/idiopathic heart failure). In fact, 123I-MIBG cardiac uptake is of prognostic value and can be used to stratify HF patients at risk for ventricular arrhythmias and sudden death. By reducing SNS hyperactivity, chronic treatment with beta-blockers improves 123I-MIBG cardiac uptake and reduces mortality in patients with HF.

Many recognizable triggers for PD appear to be associated with increased sympathetic tone, including most notably brain traumatic injuries, but also microbiota perturbations, air pollution, heavy metals like iron and manganese, and finally aging itself. In addition, there is reason to believe that SNS overactivity might trigger the principal pre-motor symptoms of PD, including hyposmia, constipation and RBD. Finally, SNS overactivity typically drives reduced low-frequency heart rate variability (HRV), another clinical sign associated with pre-motor - particularly RBD - and early PD. Interestingly, low delayed uptake and high washout rate, the 123I-MIBG scintigraphy indices of increased adrenergic drive, are typically described in PD patients.

Based on these considerations, the investigators hypothesize that 123I-MIBG cardiac impairment in neurodegenerative disease shares the same pathophysiology of other chronic conditions like HF, at least in the very early, pre-motor stages of development. Therefore, treatment of SNS hyperactivity with adrenergic blockers will improve cardiac sympathetic denervation in PD patients, providing evidence that this process is reversible. If this is true, the early detection of 123I-MIBG cardiac impairment in PD, particularly in the pre-motor phase, might create a considerable window of opportunity for treatment with adrenergic blockers - or similar compounds able to reduce SNS hyperactivity - which may result in long-term benefit such as delaying the neurodegenerative process and the onset of neurological symptoms. This may be documented and monitored using nigrostriatal dopaminergic scintigraphy (DAT scan), a strategy that would implement a dual imaging algorithm to provide early and viable biomarkers of the neurodegenerative process.

Among adrenergic blockers, carvedilol is particularly well-suited to block impaired sympathetic over-activation in virtue of several effects on the adrenoceptors, including β-1 and β-2 adrenergic blockade and α-1 adrenergic blockade, in addition to antioxidant activity, L-type calcium channel blockade, and inhibition of stress-activated protein kinase. Absorption of current oral formulations of carvedilol is typically rapid and complete, with an average elimination half -life of about 8 hours. The high lipophilic structure of carvedilol makes it one of the beta-blockers most readily crossing the blood brain barrier. Carvedilol is associated with greater reduction of sympathetic activity, as measured by 123I-MIBG myocardial uptake, than metoprolol and other selective beta-blockers. In addition, due to its α-1 adrenergic blockade properties, carvedilol may exert beneficial effects on olfactory dysfunction and insulin resistance, two abnormalities frequently associated with the neurodegenerative process in PD. Adrenergic blockers have been associated with sleep disturbances including RBD, although the latter is based on isolated anecdotal reports. The negative effect of beta-blockers on sleep quality and duration appears to be related with the suppression of night time levels of melatonin. Interestingly however, carvedilol is not associated with melatonin suppression.

The purpose of this pilot study is to investigate the effect of treatment with the adrenergic blocker carvedilol on 123I-MIBG myocardial uptake in a population of subjects with defined pre-motor PD risks (i.e. hyposmia and RBD) and abnormal baseline 123I-MIBG uptake, with or without 123I-Ioflupane uptake abnormality or PD motor symptoms. Scintigraphic changes will be correlated to motor and non-motor severity of PD, measured by validated clinical scales and cardiac autonomic function tests.

ELIGIBILITY:
Inclusion Criteria:

Male or female of age between 50 and 85 years at time of enrollment.

Diagnosis of idiopathic REM sleep behavior disorder (iRBD) or Diagnosis of hyposmia. Diagnosis of RBD will be, established either as 'definite RBD' according to the criteria proposed by the International Classification of Sleep Disorders (ICSD)-2 [AASM, 2005] or 'probable RBD' following a score of 6 or higher in the RBD questionnaire (RBDSQ) with a score of at least 1 in subitems 6.1 to 6.4 of question 6.

At least one of the following:

1. Diagnosis of hyposmia. Diagnosis of hyposmia will be established as a University of Pennsylvania Smell Identification Test (UPSIT) score < 20th percentile for the individual's age group and sex.
2. Functional constipation, assessed by a scores > 4 on a questionnaire based on modified ROME III diagnostic criteria.
3. Color vision abnormality, as assessed using HRR Pseudoisochromatic Plates, in the absence of congenital dyschromatopsia.
4. Symptoms of depression, as assessed by a Beck Depression Inventory (BDI) fast screen score >3 or concurrent use of antidepressant medications

   * Abnormal 123I-MIBG myocardial scintigraphy, as defined by a Late H/M ratio < 2.2 and/or a WR >30%, with normal cardiac ejection fraction (LVEF >55%).
   * Capacity to give informed consent

Exclusion Criteria:

Secondary Parkinsonism, including tardive

Concurrent dementia defined by a score lower than 22 on the MoCA

Concurrent severe depression defined by a BDI fast screen score greater than 13

Comorbidities related to SNS hyperactivity

Heart failure (LVEF <45%)

Recent myocardial revascularization (<12 weeks)

Chronic Hypertension (SBP>140mmHg-DBP>90mmHg)

Atrial fibrillation

Diabetes mellitus

COPD

Sleep Apnea

Severely reduced kidney function (Glomerular Filtration Rate<30ml/min)

Contraindications to the use of carvedilol

Asthma or bronchospasm

Recent myocardial infarction (<48 h)

Ongoing unstable angina

Cardiogenic shock or prolonged hypotension

Second or Third-Degree AV block

Significant valvular aortic stenosis

Obstructive cardiomyopathy, or constrictive pericarditis

Symptomatic Bradycardia (HR<60) or Sick Sinus Syndrome

Stroke within the past 1 month

Severe Hepatic Dysfunction

Allergy/hypersensitivity to iodine or study medication

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-04-04 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
123I-MIBG reuptake changes | At baseline and at 26 weeks of treatment.
  123I-MIBG reuptake will be measured by early and late Heart to Mediastinal ratio (H/M) and Washout ratio (WR) which will be calculated using the following formula: [(early heart counts/pixel - early mediastinum counts/pixel) - (late heart counts/pixel decay-corrected - late mediastinum counts/pixel decay-corrected)]/(early heart counts/pixel - early mediastinum counts/pixel). Care will be taken to exclude lung or liver from the myocardial and large vessels and lung from the mediastinum region of interest. MIBG abnormality cutoffs will be set for values of late H/M <2.2 and WR >30%.

SECONDARY OUTCOMES:
Adverse Events frequency | every 3 months up to 34 weeks
  Safety will be monitored collecting the type and frequency of adverse events, including clinical symptoms, changes in vital signs, clinical laboratory measures and EKG abnormalities.
Heart rate variability changes | At baseline and at 26 weeks of treatment.
  Twenty-four-hour Holter monitoring of all patients will be conducted at two points during the study: 1) After MIBG and prior to the administration of the study drug and 2) within one week of the end of the six-month treatment trial. Two-channel Holter recordings will obtained and analyzed on a commercially available scanner in the cardiac laboratory at Cedars Sinai Medical Center, according to published guidelines.

OTHER OUTCOMES:
MDS-UPDRS part III changes | At baseline and at 26 weeks of treatment.
  The Movement disorder society-unified Parkinson's disease rating scale (MDS-UPDRS) Part III will be administered at baseline and 26 weeks after study medication titration. Each item of the MDS-UPDRS has a possible rating from 0 to 4, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe.Clinical scales will be performed OFF medication in those subjects that might be receiving dopaminergic drugs
Sleep changes as measured by REM Behavior Disorder questionnaire | At baseline and at 26 weeks of treatment.
  RBD questionnaire (RBDSQ) changes from Screening at 26 weeks after study drug titration
Smell changes as measured by University of Pennsylvania Smell Identification Test (UPSIT) | At baseline and at 26 weeks of treatment.
  University of Pennsylvania Smell Identification Test (UPSIT) changes from screening at 26 weeks after study medication titration
Constipation score changes using a questionnaire based on modified ROME III diagnostic criteria | At baseline and at 26 weeks of treatment.
  Functional constipation will be assessed at screening and at 26 weeks after study medication titration using a questionnaire based on modified ROME III diagnostic criteria, which focuses on symptoms including straining, lumpy or hard stools, sensation of incomplete evacuation, sensation of anorectal obstruction or blockage, manual maneuvers to facilitate evacuation, and two or fewer bowel movements per week. This questionnaire is based on a six item self-report measures with a three point summated rating scale. The total score has a range of 0 to 12, with scores > 4 identifying functional constipation.
Color vision changes as measured by HRR Pseudochromatic Plates | At baseline and at 26 weeks of treatment.
  Color vision changes will be assessed using HRR Pseudochromatic Plates from screening at 26 weeks after study medication titration
DAT scan Changes | At baseline and at 26 weeks of treatment.
  DaT/SPECT uptake at baseline will be quantified at baseline and 26 weeks after study medication titration
Non-Motor Symptoms Scale (NMSS) changes | At baseline and at 26 weeks of treatment.
  The NMSS measures non-motor symptoms over the previous month. Each symptom is scored with respect to: Severity: 0 = None, 1 = Mild; 2 = Moderate; 3 = Severe and Frequency: 1 = Rarely (<1/wk); 2 = Often (1/wk); 3 = Frequent (several times per week); 4 = Very Frequent (daily or all the time).
Scopa-AUT changes | At baseline and at 26 weeks of treatment.
  The SCOPA-AUT scale consists of 25 items assessing autonomic symptoms in the following regions: gastrointestinal (7), urinary (6), cardiovascular (3), thermoregulatory (4), pupillomotor (1), and sexual (2 items for men and 2 items for women) dysfunction.
Peripheral insulin resistance changes | At baseline and at 26 weeks of treatment.
  Peripheral IR will be defined by testing for fasting plasma insulin (FPI), fasting plasma glucose (FPG) and glycated hemoglobin (HbA1c) from baseline at 26 weeks after study medication titration. HOMA index will be calculated by the formula: HOMA-IR = (FPI x FPG)/405. [A cutoff HOMA index of 2.0, equivalent to <50% sensitivity, will be used to define IR. Subjects were considered to have IR if they either had a HOMA≥2.0 and/or HbA1c≥5.7.
Central insulin resistance changes | At baseline and at 26 weeks of treatment.
  Measures of insulin sensitivity in neuronal-origin enriched plasma EVs (central IR) will be used to test the association of changes in such sensitivity to changes in MIBG uptake and clinical scores from baseline to 26 weeks after carvedilol titration. For that purpose, plasma samples will be collected and stored and -80oC to allow for isolation of neuronal origin EVs at the completion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tagliati, MD, FAAN, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Michele L Lima Gregorio, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amino T, Orimo S, Itoh Y, Takahashi A, Uchihara T, Mizusawa H. Profound cardiac sympathetic denervation occurs in Parkinson disease. Brain Pathol. 2005 Jan;15(1):29-34. doi: 10.1111/j.1750-3639.2005.tb00097.x. PMID 15779234
- [Background] Boeve BF. REM sleep behavior disorder: Updated review of the core features, the REM sleep behavior disorder-neurodegenerative disease association, evolving concepts, controversies, and future directions. Ann N Y Acad Sci. 2010 Jan;1184:15-54. doi: 10.1111/j.1749-6632.2009.05115.x. PMID 20146689
- [Background] Braak H, Del Tredici K, Rub U, de Vos RA, Jansen Steur EN, Braak E. Staging of brain pathology related to sporadic Parkinson's disease. Neurobiol Aging. 2003 Mar-Apr;24(2):197-211. doi: 10.1016/s0197-4580(02)00065-9. PMID 12498954
- [Background] Bugalho P, Mendonca M, Lampreia T, Miguel R, Barbosa R, Salavisa M. Heart rate variability in Parkinson disease and idiopathic REM sleep behavior disorder. Clin Auton Res. 2018 Dec;28(6):557-564. doi: 10.1007/s10286-018-0557-4. Epub 2018 Aug 20. PMID 30128681
- [Background] de Milliano PA, van Eck-Smit BL, de Groot AC, Lie KI. Metoprolol-induced changes in myocardial (123)I-metaiodobenzylguanidine uptake in Parkinson's disease. Circulation. 2000 Nov 14;102(20):2553-4. doi: 10.1161/01.cir.102.20.2553. No abstract available. PMID 11076832
- [Background] de Peuter OR, Verberne HJ, Kok WE, van den Bogaard B, Schaap MC, Nieuwland R, Meijers JC, Somsen GA, Bakx A, Kamphuisen PW. Differential effects of nonselective versus selective beta-blockers on cardiac sympathetic activity and hemostasis in patients with heart failure. J Nucl Med. 2013 Oct;54(10):1733-9. doi: 10.2967/jnumed.113.120477. Epub 2013 Aug 22. PMID 23970363
- [Background] Dinan TG, Cryan JF. Regulation of the stress response by the gut microbiota: implications for psychoneuroendocrinology. Psychoneuroendocrinology. 2012 Sep;37(9):1369-78. doi: 10.1016/j.psyneuen.2012.03.007. Epub 2012 Apr 5. PMID 22483040
- [Background] Dorschner J, Farmakis G, Behnke S, Hellwig D, Schneider S, Fassbender K, Kirsch CM, Dillmann U, Spiegel J. Myocardial MIBG scintigraphy may predict the course of motor symptoms in Parkinson's disease. Parkinsonism Relat Disord. 2011 Jun;17(5):372-5. doi: 10.1016/j.parkreldis.2011.03.001. Epub 2011 Mar 21. PMID 21421334
- [Background] Fereshtehnejad SM, Montplaisir JY, Pelletier A, Gagnon JF, Berg D, Postuma RB. Validation of the MDS research criteria for prodromal Parkinson's disease: Longitudinal assessment in a REM sleep behavior disorder (RBD) cohort. Mov Disord. 2017 Jun;32(6):865-873. doi: 10.1002/mds.26989. Epub 2017 Apr 21. PMID 28429825
- [Background] Goldstein DS, Holmes C, Li ST, Bruce S, Metman LV, Cannon RO 3rd. Cardiac sympathetic denervation in Parkinson disease. Ann Intern Med. 2000 Sep 5;133(5):338-47. doi: 10.7326/0003-4819-133-5-200009050-00009. PMID 10979878
- [Background] Halsband C, Zapf A, Sixel-Doring F, Trenkwalder C, Mollenhauer B. The REM Sleep Behavior Disorder Screening Questionnaire is not Valid in De Novo Parkinson's Disease. Mov Disord Clin Pract. 2018 Mar 1;5(2):171-176. doi: 10.1002/mdc3.12591. eCollection 2018 Mar-Apr. PMID 30009211
- [Background] He SC, Niu Q. Subclinical neurophysiological effects of manganese in welding workers. Int J Immunopathol Pharmacol. 2004 May-Aug;17(2 Suppl):11-6. doi: 10.1177/03946320040170S203. PMID 15345186
- [Background] Heffernan DS, Inaba K, Arbabi S, Cotton BA. Sympathetic hyperactivity after traumatic brain injury and the role of beta-blocker therapy. J Trauma. 2010 Dec;69(6):1602-9. doi: 10.1097/TA.0b013e3181f2d3e8. No abstract available. PMID 21045744
- [Background] Hogg E, Athreya K, Basile C, Tan EE, Kaminski J, Tagliati M. High Prevalence of Undiagnosed Insulin Resistance in Non-Diabetic Subjects with Parkinson's Disease. J Parkinsons Dis. 2018;8(2):259-265. doi: 10.3233/JPD-181305. PMID 29614702
- [Background] Iranzo A, Santamaria J. Bisoprolol-induced rapid eye movement sleep behavior disorder. Am J Med. 1999 Oct;107(4):390-2. doi: 10.1016/s0002-9343(99)00245-4. No abstract available. PMID 10527042
- [Background] Iwanaga K, Wakabayashi K, Yoshimoto M, Tomita I, Satoh H, Takashima H, Satoh A, Seto M, Tsujihata M, Takahashi H. Lewy body-type degeneration in cardiac plexus in Parkinson's and incidental Lewy body diseases. Neurology. 1999 Apr 12;52(6):1269-71. doi: 10.1212/wnl.52.6.1269. PMID 10214756
- [Background] Jacob S, Rett K, Wicklmayr M, Agrawal B, Augustin HJ, Dietze GJ. Differential effect of chronic treatment with two beta-blocking agents on insulin sensitivity: the carvedilol-metoprolol study. J Hypertens. 1996 Apr;14(4):489-94. PMID 8761899
- [Background] Jacobson AF, Senior R, Cerqueira MD, Wong ND, Thomas GS, Lopez VA, Agostini D, Weiland F, Chandna H, Narula J; ADMIRE-HF Investigators. Myocardial iodine-123 meta-iodobenzylguanidine imaging and cardiac events in heart failure. Results of the prospective ADMIRE-HF (AdreView Myocardial Imaging for Risk Evaluation in Heart Failure) study. J Am Coll Cardiol. 2010 May 18;55(20):2212-21. doi: 10.1016/j.jacc.2010.01.014. Epub 2010 Feb 25. PMID 20188504
- [Background] Johnson ME, Stecher B, Labrie V, Brundin L, Brundin P. Triggers, Facilitators, and Aggravators: Redefining Parkinson's Disease Pathogenesis. Trends Neurosci. 2019 Jan;42(1):4-13. doi: 10.1016/j.tins.2018.09.007. Epub 2018 Oct 17. PMID 30342839
- [Background] Joyner MJ, Barnes JN, Hart EC, Wallin BG, Charkoudian N. Neural control of the circulation: how sex and age differences interact in humans. Compr Physiol. 2015 Jan;5(1):193-215. doi: 10.1002/cphy.c140005. PMID 25589269
- [Background] Keating GM, Jarvis B. Carvedilol: a review of its use in chronic heart failure. Drugs. 2003;63(16):1697-741. doi: 10.2165/00003495-200363160-00006. PMID 12904089
- [Background] Langston JW, Wiley JC, Tagliati M. Optimizing Parkinson's disease diagnosis: the role of a dual nuclear imaging algorithm. NPJ Parkinsons Dis. 2018 Feb 23;4:5. doi: 10.1038/s41531-018-0041-9. eCollection 2018. PMID 29507872
- [Background] Lotsch J, Daiker H, Hahner A, Ultsch A, Hummel T. Drug-target based cross-sectional analysis of olfactory drug effects. Eur J Clin Pharmacol. 2015 Apr;71(4):461-71. doi: 10.1007/s00228-015-1814-2. Epub 2015 Feb 11. PMID 25666029
- [Background] Marek KL, Seibyl JP, Zoghbi SS, Zea-Ponce Y, Baldwin RM, Fussell B, Charney DS, van Dyck C, Hoffer PB, Innis RP. [123I] beta-CIT/SPECT imaging demonstrates bilateral loss of dopamine transporters in hemi-Parkinson's disease. Neurology. 1996 Jan;46(1):231-7. doi: 10.1212/wnl.46.1.231. PMID 8559382
- [Background] Martinelli N, Olivieri O, Girelli D. Air particulate matter and cardiovascular disease: a narrative review. Eur J Intern Med. 2013 Jun;24(4):295-302. doi: 10.1016/j.ejim.2013.04.001. Epub 2013 May 4. PMID 23647842
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Mitsui J, Saito Y, Momose T, Shimizu J, Arai N, Shibahara J, Ugawa Y, Kanazawa I, Tsuji S, Murayama S. Pathology of the sympathetic nervous system corresponding to the decreased cardiac uptake in 123I-metaiodobenzylguanidine (MIBG) scintigraphy in a patient with Parkinson disease. J Neurol Sci. 2006 Apr 15;243(1-2):101-4. doi: 10.1016/j.jns.2005.11.034. Epub 2006 Jan 27. PMID 16442563
- [Background] Miyamoto T, Miyamoto M, Inoue Y, Usui Y, Suzuki K, Hirata K. Reduced cardiac 123I-MIBG scintigraphy in idiopathic REM sleep behavior disorder. Neurology. 2006 Dec 26;67(12):2236-8. doi: 10.1212/01.wnl.0000249313.25627.2e. PMID 17190953
- [Background] Mizutani Y, Nakamura T, Okada A, Suzuki J, Watanabe H, Hirayama M, Sobue G. Hyposmia and cardiovascular dysautonomia correlatively appear in early-stage Parkinson's disease. Parkinsonism Relat Disord. 2014 May;20(5):520-4. doi: 10.1016/j.parkreldis.2014.02.010. Epub 2014 Feb 20. PMID 24637128
- [Background] Morrison I, Frangulyan R, Riha RL. Beta-blockers as a cause of violent rapid eye movement sleep behavior disorder: a poorly recognized but common cause of violent parasomnias. Am J Med. 2011 Jan;124(1):e11. doi: 10.1016/j.amjmed.2010.04.023. Epub 2010 Sep 29. No abstract available. PMID 20887968
- [Background] Nakajo M, Shapiro B, Glowniak J, Sisson JC, Beierwaltes WH. Inverse relationship between cardiac accumulation of meta-[131I]iodobenzylguanidine (I-131 MIBG) and circulating catecholamines in suspected pheochromocytoma. J Nucl Med. 1983 Dec;24(12):1127-34. PMID 6644373
- [Background] Searles Nielsen S, Gross A, Camacho-Soto A, Willis AW, Racette BA. beta2-adrenoreceptor medications and risk of Parkinson disease. Ann Neurol. 2018 Nov;84(5):683-693. doi: 10.1002/ana.25341. Epub 2018 Oct 30. PMID 30225948
- [Background] Nomura T, Inoue Y, Kagimura T, Uemura Y, Nakashima K. Utility of the REM sleep behavior disorder screening questionnaire (RBDSQ) in Parkinson's disease patients. Sleep Med. 2011 Aug;12(7):711-3. doi: 10.1016/j.sleep.2011.01.015. Epub 2011 Jun 22. PMID 21700495
- [Background] Nul D, Zambrano C, Diaz A, Ferrante D, Varini S, Soifer S, Grancelli H, Doval H; Grupo de Estudio de la Sobrevida en la Insuficiencia Cardiaca en Argentina. Impact of a standardized titration protocol with carvedilol in heart failure: safety, tolerability, and efficacy-a report from the GESICA registry. Cardiovasc Drugs Ther. 2005 Mar;19(2):125-34. doi: 10.1007/s10557-005-1497-5. PMID 16025231
- [Background] Orimo S, Ozawa E, Nakade S, Sugimoto T, Mizusawa H. (123)I-metaiodobenzylguanidine myocardial scintigraphy in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1999 Aug;67(2):189-94. doi: 10.1136/jnnp.67.2.189. PMID 10406987
- [Background] Orimo S, Uchihara T, Nakamura A, Mori F, Kakita A, Wakabayashi K, Takahashi H. Axonal alpha-synuclein aggregates herald centripetal degeneration of cardiac sympathetic nerve in Parkinson's disease. Brain. 2008 Mar;131(Pt 3):642-50. doi: 10.1093/brain/awm302. Epub 2007 Dec 13. PMID 18079166
- [Background] Orimo S, Suzuki M, Inaba A, Mizusawa H. 123I-MIBG myocardial scintigraphy for differentiating Parkinson's disease from other neurodegenerative parkinsonism: a systematic review and meta-analysis. Parkinsonism Relat Disord. 2012 Jun;18(5):494-500. doi: 10.1016/j.parkreldis.2012.01.009. Epub 2012 Feb 8. PMID 22321865
- [Background] Otsuka N, Ohi M, Chin K, Kita H, Noguchi T, Hata T, Nohara R, Hosokawa R, Fujita M, Kuno K. Assessment of cardiac sympathetic function with iodine-123-MIBG imaging in obstructive sleep apnea syndrome. J Nucl Med. 1997 Apr;38(4):567-72. PMID 9098203
- [Background] Packer M, Bristow MR, Cohn JN, Colucci WS, Fowler MB, Gilbert EM, Shusterman NH. The effect of carvedilol on morbidity and mortality in patients with chronic heart failure. U.S. Carvedilol Heart Failure Study Group. N Engl J Med. 1996 May 23;334(21):1349-55. doi: 10.1056/NEJM199605233342101. PMID 8614419
- [Background] Pagano G, Tan EE, Haider JM, Bautista A, Tagliati M. Constipation is reduced by beta-blockers and increased by dopaminergic medications in Parkinson's disease. Parkinsonism Relat Disord. 2015 Feb;21(2):120-5. doi: 10.1016/j.parkreldis.2014.11.015. Epub 2014 Nov 25. PMID 25483722
- [Background] Postuma RB, Montplaisir J, Lanfranchi P, Blais H, Rompre S, Colombo R, Gagnon JF. Cardiac autonomic denervation in Parkinson's disease is linked to REM sleep behavior disorder. Mov Disord. 2011 Jul;26(8):1529-33. doi: 10.1002/mds.23677. Epub 2011 Apr 29. PMID 21538520
- [Background] Sakakibara R, Tateno F, Kishi M, Tsuyusaki Y, Terada H, Inaoka T. MIBG myocardial scintigraphy in pre-motor Parkinson's disease: a review. Parkinsonism Relat Disord. 2014 Mar;20(3):267-73. doi: 10.1016/j.parkreldis.2013.11.001. Epub 2013 Nov 21. PMID 24332912
- [Background] Sakata K, Shirotani M, Yoshida H, Kurata C. Cardiac sympathetic nervous system in early essential hypertension assessed by 123I-MIBG. J Nucl Med. 1999 Jan;40(1):6-11. PMID 9935049
- [Background] Scheer FA, Morris CJ, Garcia JI, Smales C, Kelly EE, Marks J, Malhotra A, Shea SA. Repeated melatonin supplementation improves sleep in hypertensive patients treated with beta-blockers: a randomized controlled trial. Sleep. 2012 Oct 1;35(10):1395-402. doi: 10.5665/sleep.2122. PMID 23024438
- [Background] Scott LA, Kench PL. Cardiac autonomic neuropathy in the diabetic patient: does 123I-MIBG imaging have a role to play in early diagnosis? J Nucl Med Technol. 2004 Jun;32(2):66-71. PMID 15175402
- [Background] Seravalle G, Piperno A, Mariani R, Pelloni I, Facchetti R, Dell'Oro R, Cuspidi C, Mancia G, Grassi G. Alterations in sympathetic nerve traffic in genetic haemochromatosis before and after iron depletion therapy: a microneurographic study. Eur Heart J. 2016 Mar 21;37(12):988-95. doi: 10.1093/eurheartj/ehv696. Epub 2015 Dec 28. PMID 26715163
- [Background] Spiegel J, Mollers MO, Jost WH, Fuss G, Samnick S, Dillmann U, Becker G, Kirsch CM. FP-CIT and MIBG scintigraphy in early Parkinson's disease. Mov Disord. 2005 May;20(5):552-61. doi: 10.1002/mds.20369. PMID 15645531
- [Background] Spiegel J, Hellwig D, Samnick S, Jost W, Mollers MO, Fassbender K, Kirsch CM, Dillmann U. Striatal FP-CIT uptake differs in the subtypes of early Parkinson's disease. J Neural Transm (Vienna). 2007 Mar;114(3):331-5. doi: 10.1007/s00702-006-0518-2. Epub 2006 May 24. PMID 16715205
- [Background] Spiegel J, Hellwig D, Jost WH, Farmakis G, Samnick S, Fassbender K, Kirsch CM, Dillmann U. Cerebral and Extracranial Neurodegeneration are Strongly Coupled in Parkinson's Disease. Open Neurol J. 2007;1:1-4. doi: 10.2174/1874205X00701010001. Epub 2007 Aug 22. PMID 19018276
- [Background] Stoschitzky K, Koshucharova G, Lercher P, Maier R, Sakotnik A, Klein W, Liebmann PM, Lindner W. Stereoselective effects of (R)- and (S)-carvedilol in humans. Chirality. 2001 Jul;13(7):342-6. doi: 10.1002/chir.1042. PMID 11400186
- [Background] Taki J, Nakajima K, Hwang EH, Matsunari I, Komai K, Yoshita M, Sakajiri K, Tonami N. Peripheral sympathetic dysfunction in patients with Parkinson's disease without autonomic failure is heart selective and disease specific. taki@med.kanazawa-u.ac.jp. Eur J Nucl Med. 2000 May;27(5):566-73. doi: 10.1007/s002590050544. PMID 10853813
- [Background] Travin MI, Matsunari I, Thomas GS, Nakajima K, Yoshinaga K. How do we establish cardiac sympathetic nervous system imaging with 123I-mIBG in clinical practice? Perspectives and lessons from Japan and the US. J Nucl Cardiol. 2019 Aug;26(4):1434-1451. doi: 10.1007/s12350-018-1394-5. Epub 2018 Sep 3. PMID 30178272
- [Background] Treglia G, Stefanelli A, Bruno I, Giordano A. Clinical usefulness of myocardial innervation imaging using Iodine-123-meta-iodobenzylguanidine scintigraphy in evaluating the effectiveness of pharmacological treatments in patients with heart failure: an overview. Eur Rev Med Pharmacol Sci. 2013 Jan;17(1):56-68. PMID 23329524
- [Background] Valappil RA, Black JE, Broderick MJ, Carrillo O, Frenette E, Sullivan SS, Goldman SM, Tanner CM, Langston JW. Exploring the electrocardiogram as a potential tool to screen for premotor Parkinson's disease. Mov Disord. 2010 Oct 30;25(14):2296-303. doi: 10.1002/mds.23348. PMID 20976736
- [Background] Varrone A, Dickson JC, Tossici-Bolt L, Sera T, Asenbaum S, Booij J, Kapucu OL, Kluge A, Knudsen GM, Koulibaly PM, Nobili F, Pagani M, Sabri O, Vander Borght T, Van Laere K, Tatsch K. European multicentre database of healthy controls for [123I]FP-CIT SPECT (ENC-DAT): age-related effects, gender differences and evaluation of different methods of analysis. Eur J Nucl Med Mol Imaging. 2013 Jan;40(2):213-27. doi: 10.1007/s00259-012-2276-8. Epub 2012 Nov 16. PMID 23160999
- [Background] Velseboer DC, de Haan RJ, Wieling W, Goldstein DS, de Bie RM. Prevalence of orthostatic hypotension in Parkinson's disease: a systematic review and meta-analysis. Parkinsonism Relat Disord. 2011 Dec;17(10):724-9. doi: 10.1016/j.parkreldis.2011.04.016. Epub 2011 May 14. PMID 21571570
- [Background] Verberne HJ, Brewster LM, Somsen GA, van Eck-Smit BL. Prognostic value of myocardial 123I-metaiodobenzylguanidine (MIBG) parameters in patients with heart failure: a systematic review. Eur Heart J. 2008 May;29(9):1147-59. doi: 10.1093/eurheartj/ehn113. Epub 2008 Mar 17. PMID 18349024
- [Background] Wieland DM, Brown LE, Rogers WL, Worthington KC, Wu JL, Clinthorne NH, Otto CA, Swanson DP, Beierwaltes WH. Myocardial imaging with a radioiodinated norepinephrine storage analog. J Nucl Med. 1981 Jan;22(1):22-31. PMID 7452352
- [Background] Zimnik NC, Treadway T, Smith RS, Araneda RC. alpha(1A)-Adrenergic regulation of inhibition in the olfactory bulb. J Physiol. 2013 Apr 1;591(7):1631-43. doi: 10.1113/jphysiol.2012.248591. Epub 2012 Dec 24. PMID 23266935